CLINICAL TRIAL: NCT05354960
Title: Patient Reported Outcomes in Lower Limb Reconstruction in a Clinical Context
Brief Title: PROMs in Lower Limb Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nicole Lindenblatt (Other)
Responsible Party: Sponsor-Investigator, Nicole Lindenblatt, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2022-00232
Record Dates: First submitted 2022-03-16; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Patient Reported Outcome Measures; Limb Injury; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validation of LIMB-Q questionnaire: We plan to validate the questionnaires for quality of life and functional impairment in a mixed study population. In addition, CROMs, specifically the active range of motion, the 2 PD, compara-tive circumference measurements, AOFAS and MFS will be collected. In addition, photo documen-tation of the operated lower extremity will be performed. The results obtained will be correlated with each other.
  Interventions: Other: Questionnaire validation

INTERVENTIONS:
Other: Questionnaire validation — Validation and cultural adaption of the German version of the LIMB-Q

SUMMARY:
The purpose of the study is to evaluate the validity of PROMS after reconstructive surgery or amputation in the leg region. In this context, the German version of the LIMB-Q, a questionnaire-based "Patient-reported outcome measurement" (PROM), will be validated for the German-speaking region and any necessary cultural adaptations will be made for the future use of the questionnaire.

In addition, the aim is to establish a context between the LIMB-Q as a PROM and clinical outcome measurements (Maryland Foot Score, American Orthopedic Foot and Ankle Society Score).

DETAILED DESCRIPTION:
Complex tissue loss in the lower extremities is often a clinical challenge. Many different factors must be considered and weighted in the treatment algorithm, with functional restoration of the leg remaining the primary goal. Surgeon assessment alone is not sufficient to fully describe treatment outcomes. Different outcome measurement tools have been used in the past in an attempt to eval-uate these complex issues. Surgical outcomes that focus on complications and function from the physician's perspective provide valuable information but do not give a complete picture. Therefore, as in other areas of healthcare, patient-reported outcomes have become an integral part of as-sessing the quality and effectiveness of the services provided. Only a combination of clinicians' and patients' perspectives can contribute to obtaining a conclusive picture of the services provided. However, no validated patient reported outcome measure (PROM) instrument exists to date. Lower extremity injuries are life-changing events for patients. While approximately 70% undergo recon-struction, there are currently 200,0000 individuals in the United States living with a lower extremity amputation secondary to trauma. There is currently no PRO instrument in use for patients with limb-threatening lower extremity injuries. Instead, commonly used PRO instruments include the Musculoskeletal Tumor Society and the "Toronto Extremity Salvage Score", both designed for use in musculoskeletal oncology, as well as the Western Ontario and McMaster University Osteoar-thritis Index, designed for arthritis patients". These measures are limited, as they were not de-signed using qualitative interview data of patients with limb-threatening lower extremity traumatic injuries. They therefore, have not proven to be reflective of the important COI relevant to this pa-tient population. PRO instruments focusing on patients who have undergone amputation only are also in use, such as the Trinity Amputation and Prosthesis Experience Scales. However, there is no PRO instrument that is designed for all patients with limb-threatening lower extremity traumatic injuries that measures COI relevant to both reconstruction and amputation patient groups.

PRO instruments designed specifically for a given disease process are important, as they measure concepts such as satisfaction with appearance, body image, function, mobility, and psychosocial wellbeing, providing meaningful, precise, and reliable feedback on important patient- centered out-comes relevant to a specific patient population. This will allow meaningful, precise and reliable feedback on important patient-centered outcomes, with the potential for widespread use in clinical audit for quality improvement, and local, national and international research efforts.

In clinical research the LIMB-Q will have the capability to measure differences in outcomes im-portant to patients, allowing it to compare different treatments for severe lower extremity trauma. While substantial research has focused on identifying the "superior" treatment method between re-construction and amputation, this PRO instrument will be the first research instrument to allow this question to be asked while taking into account COI important to patients. In clinical care the it will provide patients with a structured and reliable method of communicating outcomes to providers, allowing for real-time adjustments in care to improve overall results.

The preliminary LIMB-Q scales have been developed using international standards for PRO in-strument development. Briefly, semi-structured qualitative interviews, combined with expert opin-ion and a literature review were used to generate a conceptual framework and preliminary set of scales. Next, cognitive debriefing interviews and solicitation of expert opinion were performed to further refine the preliminary instrument for clarity and comprehensiveness of content. The prelimi-nary LIMB-Q scales is now undergoing a large-scale, multi-institutional field test..

A comparison of outcomes assessment shows that surgeons tend to overestimate outcomes com-pared with patients. CROMs are well accepted by patients and have a high reliability. It is argued that PROM results are more difficult to interpret than objective CROMs due to higher inter- and intra-observer variability and subjective PROM assessment for cultural and other individual rea-sons. Thus, it is important to establish a context between already established CROMs and PROMs.

The purpose of the study is to evaluate the validity of PROMS after reconstructive surgery or am-putation of the legs due to trauma. The aim of the study is to validate the German version of the LIMB-Q, a questionnaire-based patient-reported outcome measurement (PROM) for the German-speaking region and to make any necessary cultural adaptations for the future use of the question-naire in order to be able to utilize the LIMB-Q in the future for all affected patients who receive re-constructive surgery or amputation of the lower extremity in the context of trauma in order to gain a better understanding of factors that have an influence on patient satisfaction. Furthermore, a con-text between the LIMB-Q as PROM and clinical outcome measures (CROMs) will be established.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients after lower extremity reconstructive surgery aged 18 years or older
* Male and female patients aged 18 years or older who have received /suffered a lower extremity amputation in the past.
* Written informed consent from the participating individual.

Exclusion Criteria:

* Patients with a tumor disease affecting the lower extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after reconstructive surgery and/or amputation of the lower extremity of the Department of Plastic Surgery and Hand Surgery, University Hospital Zurich, Switzerland
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
LIMB-Q score | 2 years
  The LIMB-Q is a new questionnaire, which has not yet been validated in German-speaking countries. It contains questions which explicitly refer to the quality of life of patients after trauma to the lower extremity who have undergone either reconstruction or amputation. The question consists of several subscales addressing different domains.
  Each question within each domain is scored from 1-4, an overall higher scores relates to higher patient satisfaction
Maryland Foot Score (MFS) | 2 years
  The Maryland Foot Score is a CROM for assessing lower extremity function. Information on pain, gait, functional limitations, aesthetics and mobility are included and scored. The maximum achievable score is 100, which corresponds to an excellent result. Gradations are made from 75-89 points (good), 60-74 points (moderate), <60 points (poor).
American Orthopedic Foot and Ankle Society Score (AOFAS) | 2 years
  The AOFAS is a clinical questionnaire that includes information from both the patient and the surgeon. The AOFAS covers four different foot regions: Ankle-Backfoot, Midfoot, Metatarsophalangeal (MTP) - Interphalangeal (IP) for the Hallux, and MTP-IP for the Little Toes. There is a separate version of the AOFAS survey for each of these four anatomical regions. Each is designed to be used independently of the others. However, each measurement consists of nine questions covering three categories: pain (40 items), function (50 items), and alignment (10 items). These are all scored together for a total of 100 points. Higher scores represent better results
Lower Extremity Functional Scale (LEFS) | 2 years
  The questionnaire contains 20 items that ask about the level of function during daily activities. The questions are answered using a 5-point Likert scale. For evaluation, the sum of the answers is calculated, whereby a maximum score of 80 can be achieved and represents an unrestricted function of the lower extremity.
Short Form- 36 (SF-36) | 2 years
  The SF-36 is a questionnaire which can be used to assess health-related quality of life. Based on 36 questions, the following qualities are evaluated: general health perception, physical health, limited physical role function, physical pain, vitality, mental health, limited emotional role function, social functioning. The possible score ranges from 0 to 100 points. 0 points represent the greatest possible restriction of health, while 100 points represent the absence of health restrictions.

SECONDARY OUTCOMES:
Active range of motion | 2 years
  The active range of motion in the knee and ankle is measured. The active range of motion in the knee is measured in the supine position with a goniometer. Active plantarflexion and dorsiflexion are measured both with the knee flexed to 90 degrees and in full extension. All measurements are compared to those of the unaffected side to calculate the deficit.
Sensitivity | 2 years
  2 point discrimination (2PD) is measured. A discrimination disk, the smallest distance that two tactile stimuli applied simultaneously to the skin must be in order to be recognized by the patient as spatially separated stimuli is measured. The 2PD is made centrally in the surgical area and at a point distal to it.
Circumference | 2 years
  Circumferential measurements are taken 10 cm above and below the knee joint, in the middle of the lower leg, at the level of the malleolus fork and at the most prominent point of the reconstruction/amputation. All measurements are compared to those of the unaffected side to calculate the deficit.
Aesthetic appearance | 2 years
  Photographic documentation of the lower limbs will allow for an assessment of the aesthetic result. It has to be taken into consideration that the first necessary condition of a judgment of taste is that it is essentially subjective. The appearance of the lower limb will be graded as good, moderate, or disagreeable by both clinicians and patients, allowing for a comparison of patient and physician experience

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Lindenblatt, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
After encryption and statistical analysis of the data, they are shared anonymously with Duke University, Durham, NC, USA using Qualtrics (www.qualtrics.com) for joint publication. At no time do the involved persons on the Duke University side have access to the original unencrypted data of the patients from the Clinic for Plastic Surgery and Hand Surgery of the University Hospital Zurich. The data will be shared to obtain a larger international study cohort for psychometric analysis and validation of the LIMB-Q.
Supporting Information: Study Protocol
Time Frame: After statistical analysis
Access Criteria: Patient data will be shared after enryption and statistical analysis

REFERENCES:
- [Background] Heidekrueger PI, Ehrl D, Prantl L, Thiha A, Weinschenk F, Forte AJ, Ninkovic M, Broer PN. Microsurgical Reconstruction of the Plantar Foot: Long-Term Functional Outcomes and Quality of Life. J Reconstr Microsurg. 2019 Jun;35(5):379-388. doi: 10.1055/s-0038-1677038. Epub 2019 Jan 9. PMID 30625504
- [Background] Kash BA, McKahan M, Tomaszewski L, McMaughan D. The four Ps of patient experience: A new strategic framework informed by theory and practice. Health Mark Q. 2018 Oct-Dec;35(4):313-325. doi: 10.1080/07359683.2018.1524598. Epub 2018 Dec 14. PMID 30551728
- [Background] Mundy LR, Grier AJ, Weissler EH, Carty MJ, Pusic AL, Hollenbeck ST, Gage MJ. Patient-reported Outcome Instruments in Lower Extremity Trauma: A Systematic Review of the Literature. Plast Reconstr Surg Glob Open. 2019 May 3;7(5):e2218. doi: 10.1097/GOX.0000000000002218. eCollection 2019 May. PMID 31333950
- [Background] Davis LA, Dandachli F, Turcotte R, Steinmetz OK. Limb-sparing surgery with vascular reconstruction for malignant lower extremity soft tissue sarcoma. J Vasc Surg. 2017 Jan;65(1):151-156. doi: 10.1016/j.jvs.2016.05.094. Epub 2016 Sep 26. PMID 27687325
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Gallagher P, MacLachlan M. Development and psychometric evaluation of the Trinity Amputation and Prosthesis Experience Scales (TAPES). Rehabil Psychol. 2000;45(2):130-154. doi:10.1037/0090-5550.45.2.130
- [Background] Mundy LR, Klassen A, Grier J, Carty MJ, Pusic AL, Hollenbeck ST, Gage MJ. Development of a Patient-Reported Outcome Instrument for Patients With Severe Lower Extremity Trauma (LIMB-Q): Protocol for a Multiphase Mixed Methods Study. JMIR Res Protoc. 2019 Oct 17;8(10):e14397. doi: 10.2196/14397. PMID 31625944
- [Background] Mundy LR, Klassen A, Sergesketter AR, Grier AJ, Carty MJ, Hollenbeck ST, Pusic AL, Gage MJ. Content Validity of the LIMB-Q: A Patient-Reported Outcome Instrument for Lower Extremity Trauma Patients. J Reconstr Microsurg. 2020 Nov;36(9):625-633. doi: 10.1055/s-0040-1713669. Epub 2020 Jul 2. PMID 32615610
- [Background] Janssen SJ, van Rein EA, Paulino Pereira NR, Raskin KA, Ferrone ML, Hornicek FJ, Lozano-Calderon SA, Schwab JH. The Discrepancy between Patient and Clinician Reported Function in Extremity Bone Metastases. Sarcoma. 2016;2016:1014248. doi: 10.1155/2016/1014248. Epub 2016 Sep 20. PMID 27725792
- [Background] Joswig H, Stienen MN, Smoll NR, Corniola MV, Chau I, Schaller K, Hildebrandt G, Gautschi OP. Patients' Preference of the Timed Up and Go Test or Patient-Reported Outcome Measures Before and After Surgery for Lumbar Degenerative Disk Disease. World Neurosurg. 2017 Mar;99:26-30. doi: 10.1016/j.wneu.2016.11.039. Epub 2016 Nov 29. PMID 27913260
- [Background] Gautschi OP, Corniola MV, Schaller K, Smoll NR, Stienen MN. The need for an objective outcome measurement in spine surgery--the timed-up-and-go test. Spine J. 2014 Oct 1;14(10):2521-2. doi: 10.1016/j.spinee.2014.05.004. No abstract available. PMID 25256899
- [Background] SooHoo NF, Vyas R, Samimi D. Responsiveness of the foot function index, AOFAS clinical rating systems, and SF-36 after foot and ankle surgery. Foot Ankle Int. 2006 Nov;27(11):930-4. doi: 10.1177/107110070602701111. PMID 17144955
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Maryland Foot Score. J Orthop Trauma. 2006;20(8). https://journals.lww.com/jorthotrauma/Fulltext/2006/09001/Maryland_Foot_Score.22.as